CLINICAL TRIAL: NCT03714698
Title: Effects of Pilates-based Exercises on Functional Capacity and Mental Health in Patients With Schizophrenia
Brief Title: Effects of Pilates Exercise Program in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gizem Irem KINIKLI, Associate Professor, PhD., PT, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2015-84-21/10
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Pilates exercise
MeSH Terms: conditions — Schizophrenia | interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: Pilates exercise group participated in supervised Pilates-based group training twice per week for six weeks, while the control group participated in a routine non-specific activity program twice a week in Community Mental Health Center during study
Who Masked: Participant, Outcomes Assessor
Masking Description: Both groups received the similar medication (atypical antipsychotic drugs) during the study. Patients in the control group participated in a non-specific activity programme including conventional exercise training, hobby and social interaction activities routinely twice a week, at the community mental health center during six weeks. The PEG participated in a supervised Pilates exercise program twice per week for six weeks (totally 12 sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Exercise Group (Active Comparator): Pilates exercise group participated in supervised Pilates-based group training twice per week for six weeks
  Interventions: Other: Pilates exercise group
- Control Group (Placebo Comparator): the control group participated in a routine non-specific activity program twice a week in Community Mental Health Center during study
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Pilates exercise group — Pilates exercise group participated in supervised Pilates-based group training twice per week for six weeks
  Other Names: non-specific; activity; program
  Arms: Pilates Exercise Group
Other: Control Group — The control group participated in a routine non-specific activity program twice a week in Community Mental Health Center during study
  Arms: Control Group

SUMMARY:
Schizophrenia is one of the most frequent psychiatric disorders with a prevalence of 0.5-1.0 % all over the world. It remains one of the major reasons for disability although medical and psychosocial interventions.

People suffering from schizophrenia may also have many complex health troubles such as cardiovascular disease, metabolic disease, diabetes mellitus, and pulmonary problems.

Researchers have been debating the utility of exercise over depression, anxiety, and obsessive-compulsive symptoms last decades. Studies indicate that physical activity improves mood, self-esteem, energy, motivation, concentration, cognitive skills, quality of life, and social interactions. Particularly in the last decade studies have been carried out showing that various exercise approaches and physical activities contribute positively to the physical and mental health of schizophrenic patients. Clinic impacts of these interventions, dominantly including aerobic exercise, strengthening and fitness training, also varied according to the type, duration and intensity of the method used.

The knowledge obtained about schizophrenia patients point out that physically and mentally holistic approaches should be required to this complicated disease. Previous trials demonstrated that various physical activity or exercise methods have positive effects in patients with schizophrenia. However, to the best of the our knowledge, literature lacks investigation about benefits of Pilates on several domains, in particular about the potential changes on physical and mental health in patients with schizophrenia. The aim of this study was to investigate the effects of Pilates-based exercise training on the physical and mental health of schizophrenia patients.

DETAILED DESCRIPTION:
Pilates exercises developed by Joseph Pilates has an increasing popularity in last decades. Pilates supposed that the balance between body and mind is an important factor in achieving health and happiness. Pilates stimulates the mind and decreases mental strain. The basic principles of Pilates-based approach are concentration, control, centering, diaphragmatic breathing, lightness, precision, and relaxation. It also aims to enlighten the awareness of body by inducing mind control. The control of large group muscles with coordination and focusing on breathing may increase aerobic capacity, and further improves mental health. Heretofore, some researchers also reported that the holistic approach of Pilates-based training may provide physical and psychological improvements on human health, and various intensities benefit the quality of life, mental health, physical fitness levels, and body types. Pilates exercises are utilized with a wide range spectrum for many diseases' management and are particularly used also for mental health disease such as depression, anxiety, mood etc. The sample of the study consisted of patients who were diagnosed with schizophrenia according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Current study was conducted in accordance with the Helsinki Declaration and its subsequent amendments. All the subjects volunteered to participate in this research and signed the informed consent form approved by the Institutional Clinical Research Ethics Committee (Protocol no: 2015-84-21/10). On receipt of a completed consent form, patients were assigned to Pilates exercise group (PEG) or control group (CG) based on their willingness.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were having symptoms of schizophrenia for at least six months, not to change the type of antipsychotic medication prescribed for at least six weeks prior to study (although dosage might change).

Exclusion Criteria:

* Patients with a severe physical disability or a physical condition that makes their participation impossible or potentially harmful (such as serious musculoskeletal or neurological disabilities) were excluded from the study. Additionally, patients who did not attend at least 10 of the 12 training sessions in the study group were excluded from the study.

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline "6 Minute Walk Test" at 6 week | at the baseline and after six weeks
  The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. Walking is an activity performed daily by all but the most severely impaired patients. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. The self-paced 6MWT assesses the submaximal level of functional capacity. Most patients do not achieve maximal exercise capacity during the 6MWT; instead, they choose their own intensity of exercise and are allowed to stop and rest during the test.

SECONDARY OUTCOMES:
Change from baseline Calgary Depression Scale for Schizophrenia at 6 week | at the baseline and after six weeks
  The Calgary Depression Scale for Schizophrenia (CDSS) was developed to assess the level of depression in schizophrenia. It is the only depression scale designed for the assessment of depression in schizophrenia and it differentiates between depression and the negative and positive symptoms of schizophrenia. The CDSS depression score is obtained by adding each of the item scores (9 items). A score above 6 has an 82% specificity and 85% sensitivity for predicting the presence of a major depressive episode.All ratings of the items are defined according to operational criteria from 0-3.
Change from baseline The Scale for the Assessment of Negative Symptoms at 6 week | at the baseline and after six weeks
  The Scale for the Assessment of Negative Symptoms (SANS) was the first instrument developed in order to provide for comprehensive assessment of negative symptoms in schizophrenia (Andreasen, 1982, 1983). It consists of five scales that evaluate five different aspects of negative symptoms: alogia, affective blunting, avolition-apathy, anhedonia-asociality, and attentional impairment. Each of these negative symptoms can be rated globally, but in addition detailed observations are made in order to achieve the global rating.Each of the measures is defined and broken down in observable behavioral components that are rated on a 6-point scale. The rating of each of the behavioral components is followed by an item that describes the patient's subjective evaluation of the symptom as a whole.
Change from baseline The Scale for the Assessment of Positive Symptoms (SAPS) at 6 week | at the baseline and after six weeks
  The Assessment of Positive Symptoms (SAPS) permits detailed evaluation and global ratings of hallucinations, delusions, positive formal thought disorder and bizarre behaviour (Andreasen, 1984). Taken together, the two scales provide a comprehensive set of rating scales in order to measure the symptoms of schizophrenia and to assess their change over time.The scale was developed by Nancy Andreasen and was first published in 1984. SAPS is split into 4 domains, and within each domain separate symptoms are rated from 0 (absent) to 5 (severe). The scale is closely linked to the Scale for the Assessment of Negative Symptoms (SANS) which was published a few years earlier.
Change from baseline The Brief Psychiatric Rating Scale at 6 week | at the baseline and after six weeks
  The Brief Psychiatric Rating Scale (BPRS) is a rating scale which a clinician or researcher may use to measure psychiatric symptoms such as depression, anxiety, hallucinations and unusual behaviour. Each symptom is rated 1-7 and depending on the version between a total of 18-24 symptoms are scored. The scale is one of the oldest, most widely used scales to measure psychotic symptoms and was first published in 1962.The single items were rated on a seven-point scale (1, not present; 2, very mild; 3, mild; 4, moderate; 5, moderately severe; 6, severe; 7, extremely severe). Thus, the range of possible BPRS total scores is from 18 to 126.

CONTACTS AND LOCATIONS:
Overall Officials: Eda AKBAŞ, Assist.Prof., Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beebe LH, Tian L, Morris N, Goodwin A, Allen SS, Kuldau J. Effects of exercise on mental and physical health parameters of persons with schizophrenia. Issues Ment Health Nurs. 2005 Jul;26(6):661-76. doi: 10.1080/01612840590959551. PMID 16020076
- [Background] Rimes RR, de Souza Moura AM, Lamego MK, de Sa Filho AS, Manochio J, Paes F, Carta MG, Mura G, Wegner M, Budde H, Ferreira Rocha NB, Rocha J, Tavares JM, Arias-Carrion O, Nardi AE, Yuan TF, Machado S. Effects of Exercise on Physical and Mental Health, and Cognitive and Brain Functions in Schizophrenia: Clinical and Experimental Evidence. CNS Neurol Disord Drug Targets. 2015;14(10):1244-54. doi: 10.2174/1871527315666151111130659. PMID 26556069
- [Background] Oertel-Knochel V, Mehler P, Thiel C, Steinbrecher K, Malchow B, Tesky V, Ademmer K, Prvulovic D, Banzer W, Zopf Y, Schmitt A, Hansel F. Effects of aerobic exercise on cognitive performance and individual psychopathology in depressive and schizophrenia patients. Eur Arch Psychiatry Clin Neurosci. 2014 Oct;264(7):589-604. doi: 10.1007/s00406-014-0485-9. Epub 2014 Feb 2. PMID 24487666
- [Background] Firth J, Cotter J, Elliott R, French P, Yung AR. A systematic review and meta-analysis of exercise interventions in schizophrenia patients. Psychol Med. 2015 May;45(7):1343-61. doi: 10.1017/S0033291714003110. Epub 2015 Feb 4. PMID 25650668